CLINICAL TRIAL: NCT00102128
Title: Evaluation of Skeletal Myoblast Transplant for Treating Ischemic Heart Failure
Brief Title: Study to Examine the Safety and Effectiveness of Implanted Skeletal Muscle Cells (Cells Removed From the Thigh Muscle) Into Scarred Areas of Heart Muscle After Heart Attack.
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: DMC recommended stop
Sponsor: Genzyme, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SMC00202
Record Dates: First submitted 2005-01-21; First posted 2005-01-24 (Estimated); Last update posted 2015-05-22 (Estimated); Status verified 2015-05

CONDITIONS: Ischemic Heart Failure; Ischemic Heart Disease; Ischemic Cardiomyopathy
MeSH Terms: conditions — Myocardial Ischemia | interventions — Cell- and Tissue-Based Therapy

INTERVENTIONS:
Drug: Cellular Therapy (Cultured Autologous Skeletal Myoblast Transplantation)

SUMMARY:
Study to examine the safety and effectiveness of implanted skeletal muscle cells (cells removed from the thigh muscle) into scarred areas of heart muscle after heart attack.

ELIGIBILITY:
Inclusion Criteria:

* Patients recommended for coronary bypass surgery (preferably with cardiopulmonary support)
* Ejection fraction ≥15% and ≤35%
* Left ventricular myocardial infarction (MI - heart attack) ≥4 weeks prior to screening

Exclusion Criteria:

* Need for a rapid surgical coronary revascularization
* Need for any other related cardiosurgical measure during coronary surgery (e.g. mitral valve repair or valve replacement)
* Patients with a left ventricular aneurysm who is a candidate for left ventricular aneurysmectomy or left ventricular reduction surgery; patient receiving left or biventricular (BiV) pacing therapy for heart failure (unless the patient has stabilized after 6 or more months of this therapy)
* Cardiomyopathy presumed to be of non-ischemic origin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2002-11; Primary Completion 2007-04 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Recovery of contractility within previously akinetic areas of the heart (areas without motion/contraction) that have received treatment (cells from the patient's thigh muscle or placebo), and change in left ventricular EF as assessed by echocardiography

SECONDARY OUTCOMES:
Time-to-first major adverse cardiac event (cardiovascular related death, non-cardiovascular death, congestive heart failure, resuscitated sudden death, myocardial infarction (heart attack) and stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Genzyme, a Sanofi Company
Locations (28):
- Belgium (4):
  - Genzyme Corporation, Aalst
  - Genzyme Corporation, Brussels
  - Genzyme Corporation, Ghent
  - Genzyme Corporation, Leuven
- France (12):
  - Genzyme Corporation, Besançon
  - Genzyme Corporation, Bordeaux
  - Genzyme Corporation, Caen
  - Genzyme Corporation, Clermont-Ferrand
  - Genzyme Corporation, Grenoble
  - Genzyme Corporation, Lille
  - Genzyme Corporation, Lyon
  - Genzyme Corporation, Nantes
  - Genzyme Corporation, Paris
  - Genzyme Corporation, Rennes
  - Genzyme Corporation, Rouen
  - Genzyme Corporation, Toulouse
- Germany (3):
  - Genzyme Corporation, Bad Oeynhausen
  - Genzyme Corporation, Hamburg
  - Genzyme Corporation, Hanover
- Italy (5):
  - Genzyme Corporation, Bologna
  - Genzyme Corporation, Genova
  - Genzyme Corporation, Milan
  - Genzyme Corporation, Treviso
  - Genzyme Corporation, Udine
- Genzyme Corporation, Lausanne, Switzerland
- United Kingdom (3):
  - Genzyme Corporation, Cambridge
  - Genzyme Corporation, London
  - Genzyme Corporation, Southampton